CLINICAL TRIAL: NCT03584932
Title: Youth Services Navigation Intervention for HIV+ Adolescents and Young Adults Being Released From or at Risk for Incarceration: A Randomized Control Trial
Brief Title: Youth Services Navigation Intervention for HIV+ Youth Being Released From or At-risk for Incarceration
Acronym: LINK2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital Los Angeles (Other); University of Chicago (Other); Cook County Health & Hospitals System (Other)
Responsible Party: Principal Investigator, Nina T. Harawa, MPH, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MD011773-02 (NIH)
Record Dates: First submitted 2018-06-18; First posted 2018-07-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: HIV/AIDS
Keywords: Youth,; Criminal justice; Sexual/gender minorities; Navigation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Subjects participate in a youth service navigation intervention and are eligible to receive contingency management incentives.
  Interventions: Behavioral: LINK2 Youth Services Navigation Intervention
- Control arm (No Intervention): Standard of care as set forth by the national HIV care guidelines.

INTERVENTIONS:
Behavioral: LINK2 Youth Services Navigation Intervention — There will be 6 in-person sessions delivered by a youth services navigator, plus weekly check-in calls after session 2 for a total of six months. As part of the learning sessions, the participant will learn important information about HIV and how to get the most out of his/her HIV care.
  Arms: Intervention arm

SUMMARY:
HIV prevalence among incarcerated youth living with HIV (YWH) is three times that of the general population and one in seven of all persons with HIV experience incarceration each year. Furthermore, less than half of all youth in the United States with HIV achieve HIV viral load suppression, due to poor retention and adherence to anti-retroviral therapy (ART). Existing linkage and retention services are insufficient to meet the acute needs of youth with HIV who are at risk for incarceration, recently experienced incarceration or arrest, or those nearing reentry from a correctional facility. This holds particularly true in the high-need period following release from incarceration. The LINK2 study will develop and implement a youth service navigation (YSN) intervention to improve linkage and retention among YWH at risk for incarceration and with current incarceration and arrest histories and analyze results to address existing gaps in the literature.

The investigators will enroll 142 YWH, aged 16-25 (+364 days), incarcerated in Los Angeles and Chicago jails and through community providers serving those at risk for incarceration and YWH with recent incarceration and arrest histories. The investigators will randomize participants to the YSN intervention (n=71) vs. a usual-care control group (n=71). The youth services navigators (YSNs) will assist with addressing immediate unmet needs such as housing, transportation, and food prior to clinical care and ongoing; will guide intervention participants to a range of community services to support progress along the continuum of HIV care; and will provide direct ART adherence support.

The proposed study has two Primary Specific Aims:

1. Adapt an existing peer navigation intervention for adults to create a Youth Service Navigation (YSN) intervention sensitive to sexual and gender minority (SGM) culture that guides youth to needed services along the continuum of HIV care. This intervention combines medical, substance use and mental health care with comprehensive reentry support for YWH, aged 16-25 (+364 days) upon release from large county jails and juvenile detention systems or with arrests in the prior 12 months and those at risk for incarceration based on various social determinants.
2. Using a two-group RCT design, the investigators will test the effectiveness of the new YSN, youth SGM-sensitive intervention among YLWH aged 16-25 (+364 days), compared to controls offered standard of care. The investigators will evaluate the YSN Intervention's effect on post-incarceration linkage, retention, adherence, and viral suppression, as well as on substance use disorders, mental health, services utilization, and met needs. Secondary Aims: The investigators will assess YSN's effects on recidivism, costs and potential cost-offset/effectiveness.

ELIGIBILITY:
If recruited in jail:

1. Diagnosed HIV+;
2. at least 18 but younger than 26 (25 and 364 days);
3. non-cis women;
4. Fluent in speaking English;
5. Have an anticipated sentence of no more than 12 months;
6. Going to live in the State of Illinois, LA County, Kern County, San Diego County, Riverside County, Ventura County or San Bernardino County

If recruited outside of jail:

1) Diagnosed HIV+; 2) At least 16 but younger than 26 (25 and 364 days); 3) Non-cis women; 4) Fluent in speaking English; 5) Incarceration or arrest history within the last 12 months of enrollment; or 6) At risk for incarceration defined as having one or more of the following risk factors: mental illness, substance use disorder, current financial hardship, homelessness, unstable housing in the prior 6 months, foster care or parental incarceration; 7) Living in the State of Illinois, LA County, Kern County, San Diego County, Riverside County, Ventura County or San Bernardino County

Exclusion Criteria:

1. Inability to give informed consent; 2. Parole hold or transfer to prison

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Non-cis woman
Enrollment: 106 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Linkage to HIV care, retention in HIV, adherence to anti-retroviral therapy (ART), and viral suppression | 12 months
  Linkage to care HIV care is measured as HIV primary care provider visits; time to 1st post-release HIV care visit. Measures will involve survey and electronic record sources; self-reported measures derived from Outreach Initiative and HCSUS instrument. Retention in HIV care is measured as number of visits and missed visits to HIV primary care providers. Measurement tools include surveys and electronic record sources; self-reported measures derived from the Outreach Initiative and the HCSUS instrument. ART adherence is measured using a visual analogue scale of % (0-100) in surveys. Additional tools include electronic record sources; self-reported measures derived from Outreach Initiative; HCSUS instrument. Viral suppression is deemed undetectable at < 50 copies/ml as defined by the Los Angeles County Department of Public Health. Tools will include survey and electronic record sources and items from the HCSUS instrument and Outreach Initiative.

SECONDARY OUTCOMES:
Effects on recidivism, costs and potential cost-offset/effectiveness | 5 years
  Cost offsets/effectiveness will be measured as number of outpatient HIV/general primary and specialty care; number of mental health and substance abuse treatment visits and stays. Measures will involve electronic data sets for outpatient HIV primary and specialty care; and data sets for mental health and substance abuse treatment visits/stays.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No